CLINICAL TRIAL: NCT07317466
Title: Clinical Study for Precise Image for Pediatrics for Incisive CT and CT 5300 Systems
Brief Title: Precise Image for Pediatrics
Status: Not yet recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Precise Image for Pediatrics
Record Dates: First submitted 2025-09-22; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Computed Tomography
Keywords: Precise Image; CT5300; Incisive CT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this clinical study is to evaluate the performance of the Precise Image reconstruction algorithm in pediatric patients (specifically, head and body CT imaging of patients from 18 months up to and including 18 years of age). Clinical data generated from this study is intended to support a proposed expansion of the intended population of Precise Image.

The study has two objectives:

1. To evaluate the image quality and diagnostic confidence of Precise Image compared to the standard-of-care reference (iDose4) for:

   * Head and body CT images of pediatric patients (from 18 months up to and including 18 years of age).
2. To demonstrate non-inferiority of Precise Image to iDose4 for the relevant anatomy and resolution groups.

DETAILED DESCRIPTION:
This is a retrospective, observational, multi-site, controlled, blinded, non-inferiority clinical investigation.

Precise Image is a reconstruction mode using a trained deep learning neural network to generate images with reduced noise and improved low contrast detectability at lower doses compared with standard FBP (filter back projection) reconstruction.

Pediatric subjects (from 18 months up to and including 18 years of age) scanned by the FDA-cleared Philips Incisive CT (K212441) or CT 5300 (K232491) systems.

The study will include reconstructed images of 168 CT scans in total. For each of the anatomies and resolutions, 42 scans will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scanned by FDA-cleared and marketed Philips Incisive CT or CT 5300 systems, and according to the department standard of care clinical protocols for the applicable anatomies.
* Subject age: From 18 months up to and including 18 years of age.

Exclusion Criteria:

* Subject age: Below 18 months and above 18 years of age.
* Scans that were acquired using generic 'Head' and 'Body' scan types (as Precise Image does not support generic 'Head' and 'Body' scan types).
* Scans that were acquired using a kilovoltage peak of 70 kVp (as Precise Image does not support a kilovoltage peak lower than 80 kVp).
* Scans that the site radiologists have deemed as non-diagnostic image quality in standard practice (e.g. patient movement).
* Scans that are not completed due to technical difficulties.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatrics
Sampling Method: Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of CT Image quality and diagnostic confidence via 5-point Likert Scale | Reading session at 4 months
  The image quality and diagnostic confidence of Precise Image reconstructions is non-inferior to iDose4 reconstructions for head and body CT images of pediatric patients (from 18 months up to and including 18 years of age). Measurement will be done via 5-point Likert Scale for Image Quality where 5 is excellent and 1 is poor image quality.